CLINICAL TRIAL: NCT02718170
Title: Buried Intramedullary K-wire Fixation Compared With Plate and Screw Fixation in Unstable Extra-Articular Metacarpal Fractures: A Randomized, Controlled Study
Brief Title: Buried Intramedullary K-wire Fixation Compared With Plate and Screw Fixation for Metacarpal Fractures in Unstable Extra-Articular Metacarpal Fractures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00048356
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Metacarpal Fracture
MeSH Terms: interventions — Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buried Intramedullary K-wire Fixation (Experimental): Patients randomized to buried intramedullary k-wire fixation will undergo a standardized antegrade open reduction and fixation procedure with an intramedullary k-wire.
  Interventions: Procedure: Buried Intramedullary K-wire Fixation
- Plate and Screw Fixation (Active Comparator): Patients randomized to Plate and Screw Fixation will undergo a standardized open reduction and internal fixation with plate and screws. Brand of plate will be left to the operating surgeon's discretion.
  Interventions: Procedure: Plate and Screw Fixation

INTERVENTIONS:
Procedure: Buried Intramedullary K-wire Fixation
  Arms: Buried Intramedullary K-wire Fixation
Procedure: Plate and Screw Fixation
  Arms: Plate and Screw Fixation

SUMMARY:
Randomized controlled trial comparing a technique for buried intramedullary k-wire fixation to plate and screw fixation for unstable extra-articular metacarpal fractures.

DETAILED DESCRIPTION:
Metacarpal fractures are a common injury to the hand. Most fractures occur due to direct force from either a axial load to the dorsum of the metacarpophalangeal joint or low energy fall onto an outstretched hand. Many of these fractures can be treated closed with a closed reduction and splinting however, some displaced or angulated fractures require open reduction and internal fixation. Many fixation techniques have been used, however to the investigators knowledge, no one has prospectively randomized patients to compare plate and screw fixation with buried intramedullary k-wire fixation.

The purpose of this study is to compare Plate and screw and buried intramedullary fixation, using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire as the primary outcome measured. Secondary outcomes will include total active motion, complications, cost, reoperation rate.

ELIGIBILITY:
Inclusion Criteria:

* The patient has an unstable extra-articular metacarpal fracture that meets operative indications
* Informed consent is obtained from the patient or proxy
* Male or female who are 16 years of age or older

Exclusion Criteria:

* If the patients range of motion was decreased prior to injury (previous upper extremity injury, osteoarthritis, etc.)
* Pathological Fracture
* Greater than 21 days from fracture to definitive open reduction and internal fixation
* If contamination or wounds from open fractures do not permit standardized buried intramedullary fixation or plate and screw fixation
* Highly comminuted diaphyseal fractures
* Articular fractures
* Multiple fractures involving bones other than another metacarpal in the same upper extremity
* The patient had a previous upper extremity injury that has limited hand function or finger range of motion

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-03; Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Disability as measured by Disability of Arm, Shoulder and Hand Score | 3 months

SECONDARY OUTCOMES:
Total Active Motion in degrees | 3 months
  Measured by goniometer
Grip Strength | 3 months
Disability as measured by Disability of Arm, Shoulder and Hand Score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Millon, MD, Principal Investigator — Prisma Health-Upstate

IPD SHARING:
Plan to Share IPD: No